CLINICAL TRIAL: NCT01516775
Title: Untersuchung Des Magen-pH in Intubationsanästhesie Bei Kindern
Brief Title: Gastric pH in Intubated Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Achim Schmitz (Other)
Responsible Party: Sponsor-Investigator, Achim Schmitz, Principle Investigator, Consultant ("Leitender Arzt Anästhesieabteilung, Leiter Weisse Zone"), University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK-ZH Nr. 2011-0034
Record Dates: First submitted 2012-01-16; First posted 2012-01-25 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Preoperative Fasting
Keywords: preoperative care; preoperative period; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 hour fluid fasting (Experimental): allowed to drink until 1 hour before scheduled anaesthesia induction
  Interventions: Other: clear fluid ingestion
- 2 hours fluid fasting (Active Comparator): allowed to drink until 2 hour before scheduled anaesthesia induction
  Interventions: Other: clear fluid ingestion

INTERVENTIONS:
Other: clear fluid ingestion — drinking of clear fluid in preoperative period

SUMMARY:
Fasting (according to ASA, ESA or institutional guidelines) is an important strategy to minimize the risk of regurgitation, vomiting and pulmonary aspiration during general anaesthesia; the effect of fasting time for clear fluid on gastric pH in children is goal of this study and can be investigated in children undergoing elective procedures in intubation anaesthesia without inconvenience or additional invasive procedure and hence without additional risk

Hypotheses: Gastric pH is higher in children that drink until 1 hour before anaesthesia induction than in those that drink until 2 hours before anaesthesia induction

ELIGIBILITY:
Inclusion Criteria:

* age > 1 / <= 16 years
* ASA class I or II
* elective surgery requiring general anaesthesia using tracheal intubation

Exclusion Criteria:

* disease or dysfunction of gastrointestinal tract
* chronic diseases or conditions not compatible with ASA class I or II

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
gastric pH | within 10 min after tracheal intubation
  gastric pH is measured from gastric contents which is sampled in a syringe via an orogastric tube immediately during anaesthesia after tracheal intubation induction; suctioning of the stomach after intubation is a procedure routinely performed in every intubation child in our institution

SECONDARY OUTCOMES:
subjective feeling of hunger/thirst | within 10 minutes after arrival of patient in operating theatre
  subjective feeling of hunger/thirst given as rating scale from 1 to 4
gastric aspirate volume | within 10 min after tracheal intubation
  gastric aspirate volume is the amount of gastric contents which is sampled in a syringe via an orogastric tube immediately during anaesthesia after tracheal intubation induction; suctioning of the stomach after intubation is a procedure routinely performed in every intubation child in our institution
Postoperative Nausea and Vomiting (PONV) in recovery unit | recovery period, on the average within 90 minutes after end of anaesthesia
Behaviour during recovery period | recovery period, on the average within 90 minutes after end of anaesthesia
  Rating Scale 1 - 5 by blinded nurse (5: severely agitated/emergency delir with subsequent drug therapy, 4: agitated/emergeny delir; 3: slightly agitated; 2: complaining pain but cooperative; 1: cooperative)
Behaviour during anaesthesia induction | on the average within 20 minutes after arrival of patient in operating theatre
  Rating scale 1 - 5 by (blinded) anaesthetist: 1: cooperating - 2: anxious but cooperating - 3: hostile - 4: crying - 5: agitated/fighting

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Schmitz, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Schmidt AR, Buehler P, Seglias L, Stark T, Brotschi B, Renner T, Sabandal C, Klaghofer R, Weiss M, Schmitz A. Gastric pH and residual volume after 1 and 2 h fasting time for clear fluids in childrendagger. Br J Anaesth. 2015 Mar;114(3):477-82. doi: 10.1093/bja/aeu399. Epub 2014 Dec 13. PMID 25501720